CLINICAL TRIAL: NCT06913036
Title: Muscular Response to Short vs. Prolonged Cycling: A Crossover Trial on Low-Frequency Fatigue Sensitivity
Brief Title: Myocene Sensivity to Cycling Intensities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Myo_sens_001
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fatigue Intensity
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 minutes all-out (Experimental): 4 minute time trial all-out
  Interventions: Device: Low-frequency fatigue - Myocene
- 30 minute all-out (Experimental): 30 minute cycling all-out
  Interventions: Device: Low-frequency fatigue - Myocene

INTERVENTIONS:
Device: Low-frequency fatigue - Myocene — Low frequency fatigue will be measured using Myocene

SUMMARY:
This study aims to address this gap by assessing LFF following different efforts in cycling, aiming to identify a pattern. Also, we expect that this study helps to clarify to which efforts (prolonged vs short) are more likely to trigger substantial changes in LFF responses.

ELIGIBILITY:
Inclusion Criteria:

* Road cyclists

Exclusion Criteria:

* Injured or recently injured participants

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
low-frequency fatigue | Baseline, 30 minutes post, 24 hours post
  Low-frequency fatigue assessed using Myocene software, which computes the median value of the ratio between high and low frequency stimulations

IPD SHARING:
Plan to Share IPD: Undecided